CLINICAL TRIAL: NCT05376228
Title: A Systems Biology Approach for Identification of Host and Microbial Mechanisms and Druggable Targets for the Treatment of PSC-IBD
Acronym: PSC-Vanc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mohammed Nabil Quraishi, Chief Investigator and Consultant Gastroenterologist, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK7338
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Bowel Diseases; Primary Sclerosing Cholangitis
Keywords: primary sclerosing cholangitis; inflammatory bowel disease; microbiome; vancomycin
MeSH Terms: conditions — Inflammatory Bowel Diseases; Cholangitis, Sclerosing | interventions — Vancomycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Oral Vancomycin — As part of standard of care

SUMMARY:
Primary sclerosing cholangitis (PSC) is the classical hepatobiliary manifestation of inflammatory bowel disease (IBD). Although rare, PSC is associated with significant and disproportionate unmet needs; with heightened risks of colorectal cancer and colectomy, and greater all-cause mortality rates compared to matched IBD patients. Unfortunately, no medical therapy has been proven to slow disease progression in PSC-IBD, and liver transplantation is the only lifesaving intervention for patients.

The strong association between PSC and IBD has led to several pathogenic hypotheses, in which dysregulated mucosal immune responses are proposed to contribute. Of note, the investigators recently identified distinct mucosal transcriptomic profiles in PSC-IBD; with regards bile acid metabolism, bile acid signalling, and a central role of enteric dysbiosis. In parallel, pilot data from other groups have shown that treatment with oral vancomycin (a non-absorbable, gut-specific antibiotic) attenuates colonic inflammation and improves biochemical markers of cholestasis in PSC. However, there is no mechanistic data exploring the host-microbial alterations under vancomycin treatment in PSC-IBD, neither the impact of vancomycin on bile acid circulation. The investigators of this study hypothesize that oral vancomycin attenuates colonic mucosal inflammation in PSC-IBD, by restoring gut microbiota mediated bile acid homeostatic pathways. Through these means the study aims to identify druggable gut microbial and host molecular pathways associated with bile acid mediated colonic mucosal inflammation in PSC-IBD.

DETAILED DESCRIPTION:
Primary sclerosing cholangitis (PSC) is the classical hepatobiliary manifestation of inflammatory bowel disease (IBD). Although rare, PSC is associated with significant and disproportionate unmet needs; with heightened risks of colorectal cancer and colectomy, and greater all-cause mortality rates compared to age- and sex-matched IBD controls. Unfortunately, no medical therapy has been proven to slow disease progression in PSC-IBD, and liver transplantation is the only lifesaving intervention for patients. The strong association between PSC and IBD has led to several pathogenic hypotheses, in which dysregulated mucosal immune responses are proposed to contribute. Of note, the investigators of this study recently identified distinct mucosal transcriptomic profiles in PSC-IBD; with regards bile acid metabolism, bile acid signalling, and a central role of enteric dysbiosis. In parallel, pilot data from other groups have shown that treatment with oral vancomycin (a non-absorbable, gut-specific antibiotic) attenuates colonic inflammation and improves biochemical markers of cholestasis in PSC. However, there is no mechanistic data exploring the host-microbial alterations under vancomycin treatment in PSC-IBD, neither the impact of vancomycin on bile acid circulation.

In this study, fifteen PSC-IBD patients will be recruited through a large tertiary referral centre, who are undergoing lower gastrointestinal examination as per routine standard of care. Participants will be offered 4 weeks of treatment with oral vancomycin, and stool samples collected at different timepoints to evaluate changes in metagenomic, metatranscriptomic, and bile acid profiles. Colonic biopsies will be collected at baseline and at week 4 (flexible sigmoidoscopy) and subjected to FACS sorted RNA sequencing to identify changes in colonic epithelial cell pathways. Multi-omics data integration will be performed to uncover combinations of predictive profiles, model microbial networks, and host transcriptomic changes implicated in the response to oral vancomycin. This study will inform the downstream identification of specific host molecular and microbial pathways that has a potential for development of therapeutic targets for PSC-IBD in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of primary sclerosing cholangitis and concurrent colitis
* Mild to moderately active colitis based on partial Mayo score of ≥3 and ≤6
* Scheduled for a standard of care lower GI endoscopy as part of disease assessment / surveillance

Exclusion Criteria:

* History of previous colectomy
* Isolated small bowel disease
* Stricturing , fistulating or perianal phenotype
* Use of antibiotics and/or probiotics in the prior 3 months
* Use of steroids in last 2 weeks
* Commenced thiopurines / methotrexate in last 3 months
* History of intolerance to oral vancomycin
* Decompensated liver disease (Child C cirrhosis)
* Active infectious diarrhoea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 patients with active PSC-IBD will undergo 4 weeks of treatment with open label (standard of care) oral vancomycin.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Identify stool metagenomic, metatranscriptomic and bile acid profiles following treatment with oral vancomycin in PSC-IBD | 12 months
Investigate changes in colonic mucosal epithelial bile acid and immunological pathways through FACS sorted RNA-sequencing following oral vancomycin | 12 months
Identification of druggable host molecular and microbial targets through multi-omic integration analysis | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quraishi MN, Acharjee A, Beggs AD, Horniblow R, Tselepis C, Gkoutos G, Ghosh S, Rossiter AE, Loman N, van Schaik W, Withers D, Walters JRF, Hirschfield GM, Iqbal TH. A Pilot Integrative Analysis of Colonic Gene Expression, Gut Microbiota, and Immune Infiltration in Primary Sclerosing Cholangitis-Inflammatory Bowel Disease: Association of Disease With Bile Acid Pathways. J Crohns Colitis. 2020 Jul 30;14(7):935-947. doi: 10.1093/ecco-jcc/jjaa021. PMID 32016358
- [Derived] Quraishi MN, Cheesbrough J, Rimmer P, Mullish BH, Sharma N, Efstathiou E, Acharjee A, Gkoutus G, Patel A, Marchesi JR, Camuzeaux S, Chappell K, Valdivia-Garcia MA, Ferguson J, Brookes MJ, Walmsley M, Rossiter AE, van Schaik W, McInnes RS, Cooney R, Trauner M, Beggs AD, Iqbal TH, Trivedi PJ. Open Label Vancomycin in Primary Sclerosing Cholangitis-Inflammatory Bowel Disease: Improved Colonic Disease Activity and Associations With Changes in Host-Microbiome-Metabolomic Signatures. J Crohns Colitis. 2025 Feb 4;19(2):jjae189. doi: 10.1093/ecco-jcc/jjae189. PMID 39673746
- See also: Related Info — https://www.pscsupport.org.uk/vancomycin-a-promising-option-for-the-treatment-of-psc/
- See also: Related Info — https://www.pscsupport.org.uk/new-vancomycin-study-in-psc/